CLINICAL TRIAL: NCT01572623
Title: Efficacy of Two Different Pre-Intervention Therapeutic Strategies With Clopidogrel and Atorvastatin for the Prevention of Cerebral Damage During Carotid Artery Stenting. Armyda-Caro Randomized Trial.
Brief Title: Clopidogrel and Atorvastatin Treatment During Carotid Artery Stenting
Acronym: ARMYDA-CARO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Patti Giuseppe, MD, Campus Bio-Medico University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 2011-005330-18
Record Dates: First submitted 2012-04-04; First posted 2012-04-06 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Carotid Stenosis
Keywords: Therapeutic strategies for carotid artery stenting
MeSH Terms: conditions — Carotid Stenosis | interventions — Clopidogrel; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antiplatelet before carotid artery stenting (Active Comparator): Clopidogrel 600 mg after carotid artery stenting
  Interventions: Drug: Clopidogrel
- Statin therapy before carotid artery stenting (Active Comparator): Reloading dose of Atorvastatin (80 mg at 12 hours and 40 mg at 6-8 hours before carotid artery stenting) versus no reload.
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Clopidogrel — Loading dose of Clopidogrel 600 mg versus 300 mg before carotid artery stenting
  Arms: Antiplatelet before carotid artery stenting
Drug: Atorvastatin — Reloading dose of Atorvastatin (80 mg at 12 hours and 40 mg at 6-8 hours before carotid artery stenting) versus no reload.
  Arms: Statin therapy before carotid artery stenting

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of two different loading doses of Clopidogrel and a reloading of Atorvastatin in the prevention of periprocedural ischemic brain damage in patients undergoing carotid angioplasty.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic and asymptomatic patients with finding of significant carotid stenosis

Exclusion Criteria:

* patients with acute injuries to the baseline MRI of the brain,
* patients with active bleeding,
* contraindications to statin therapy and MRI contraindications (pacemaker/claustrophobic).

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Cerebral damage | 30 days
  Incidence of stroke at 30 days (defined as a neurologic deficit lasting> 24 hours with MRI evidence of cerebral ischemic injury) or transient ischemic attack (TIA);
  - Evidence of new onset acute ischemic lesions on MRI-DWI brain after the procedure, even in the absence of specific neurological symptoms

SECONDARY OUTCOMES:
Bleeding complications | 30 days
  Effect on the 30-day major and minor bleeding (according to the TIMI definition);
  - Incidence of post-procedural vascular complications (pseudoaneurysm, AV fistula, hematoma> 5 cm).

CONTACTS AND LOCATIONS:
Overall Officials: Patti Giuseppe, MD, Principal Investigator — Campus Bio-Medico University
Locations (1):
- Campus Bio Medico University of Rome, Rome, RM, Italy

REFERENCES:
- [Derived] Patti G, Tomai F, Melfi R, Ricottini E, Macri M, Sedati P, Giardina A, Aurigemma C, Leporace M, D'Ambrosio A, Di Sciascio G. Strategies of clopidogrel load and atorvastatin reload to prevent ischemic cerebral events in patients undergoing protected carotid stenting. Results of the randomized ARMYDA-9 CAROTID (Clopidogrel and Atorvastatin Treatment During Carotid Artery Stenting) study. J Am Coll Cardiol. 2013 Apr 2;61(13):1379-87. doi: 10.1016/j.jacc.2013.01.015. Epub 2013 Mar 9. PMID 23490041